CLINICAL TRIAL: NCT03443544
Title: Fournier's Gangrene and the Origin of the Infection as a Prognostic of Morbidity and Mortality, an Analysis of 121 Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Adrián Gutiérrez González, Chief of department, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: UR16-00003
Record Dates: First submitted 2018-02-12; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Fournier Gangrene; Fournier's Gangrene of Penis; Fournier's Gangrene of Scrotum
Keywords: fournier's; gangrene
MeSH Terms: conditions — Fournier Gangrene; Gangrene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Intestinal origin: Either perianal abcess or rectal carcinoma
  Interventions: Procedure: Aggressive debridement
- Testicular Origin: Complicated epididymitis with fascitis,
  Interventions: Procedure: Aggressive debridement
- Urinary Origin: From urinary tract infection or fistulae from urethral trauma
  Interventions: Procedure: Aggressive debridement
- Cutaneous Origin: mostly folliculitis, and skin infections
  Interventions: Procedure: Aggressive debridement

INTERVENTIONS:
Procedure: Aggressive debridement — Aggressive debridement of the tissues undergoing fascitis

SUMMARY:
Background:

Fournier's gangrene it's a necrotizing infection of the genital area, with high morbidity and mortality. The site of infection its the origin of the necrotizing fasciitis. There are 4 well known origins of Fournier's gangrene: Testicular, Intestinal, Urinary and cutaneous, and its prognostic value has not been established yet, that's because the lack of case series with adequate number of patients. This is a retrospective study in which we evaluate the prognostic factors of every patient and its mortality compared with its origin area and multiple scores with their survival rates and hospital stay.

DETAILED DESCRIPTION:
Objective:

To evaluate origins of Fournier's gangrene as a prognostic value in the morbidity and mortality.

Patients and methods:

This is a retrospective study where patients from a single hospital from 2007 to 2016 were included. They were categorized in 4 groups matching the origin of infection. In every group categorizing with the origin of infection and determined severity factors, days of hospital stay, Fournier's gangrene severity index and mortality. A statistic analysis will be done using lineal multivariable analysis.

ELIGIBILITY:
Inclusion Criteria

* Male Patient
* Fournier's Gangrene
* All patients treated with two antibiotics
* All patients undergone with aggressive debridement

Exclusion Criteria

* Female
* Not having Fournier's Gangrene

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male patients with Fournier's Gangrene
Study Population: Patients from a single hospital (Hospital Universitario "Dr Jose E. Gonzalez") from 2007 to 2016 were included.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Fournier's Gangrene Severity Index | 0-24 hours
  A score to predict mortality in this kind of patients
Hospital stay ( in days) | 0 to 2 months
  The patients hospital stay
Couture | 24 hours
  Positive or negative couture and the bacterias growing in the abscess

SECONDARY OUTCOMES:
Diabetes mellitus | 0 - 100 years
  if the patient had diabetes mellitus type 2 or not
Hypertension | 0 - 100 years
  if the patient had arterial hypertension or not
Alcohol drinking | 0 - 100 years
  if the patient drinks alcohol or not
Tobacco smoking | 0 - 100 years
  if the patient smokes or not

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario "Dr Jose Eleuterio Gonzalez", Monterrey, Mexico

IPD SHARING:
Plan to Share IPD: No